CLINICAL TRIAL: NCT04300842
Title: Quantifying Fatigue in Cancer Patients Using Smart Bracelet Devices
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: N201910036
Record Dates: First submitted 2019-12-22; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2019-12

CONDITIONS: Cancer-Related Condition
Keywords: Cancer-related fatigue; smart bracelet device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patient: This project expects to enroll 60 cancer patients and their subjective-objective measurements on fatigue, stress, and total steps will be observed.
  Interventions: Device: smart bracelet
- Healthy population: This project expects to enroll 60 healthy population and their subjective-objective measurements on fatigue, stress, and total steps will be observed.
  Interventions: Device: smart bracelet

INTERVENTIONS:
Device: smart bracelet — to measure the stress, fatigue, and activity.

SUMMARY:
This project expects to enroll 60 cancer patients, 60 healthy people and their subjective-objective measurements on fatigue, stress, and total steps will be validated so that the information can be used in further care and improvement of life of quality of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 20 years old;
* One group had a cancer diagnosis, one group no cancer diagnosis;
* Can continuous wearing bracelet for 5 days or more

Exclusion Criteria:

* Unclear and unable to answer the questionnaire

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer patients with some cancer treatment side effects. Healthy people compare with cancer patients who no cancer disease now.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-12-22 (Actual); Primary Completion 2020-12-26 (Estimated); Study Completion 2021-12-26 (Estimated)

PRIMARY OUTCOMES:
fatigue | over 5 days
  Unit of measure: severity of fatigue level; measurement tool: Brief Fatigue Index
Heart Rate Variability (HRV) monitor | over 5 days
  Use a digital device to measure the heart rate variability and calculate the HRV data

SECONDARY OUTCOMES:
Distress Thermometer(DT) | over 5 days
  a screening measure to identify and address psychological distress in individuals with cancer. a cutoff score of 3 on the DT to indicate patients with clinically elevated levels of distress.
Leeds Sleep Evaluation Questionnaire(LSEQ） | over 5 days
  To assess sleep quality, higher scores mean more disrupt sleep.
International Physical Activity Questionnaire(IPAQ） | over 5 days
  Life activity survey
Perceived Stress Scale (PSS） | over 5 days
  higher scores mean more stressful condition

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes